CLINICAL TRIAL: NCT05400226
Title: A Phase 2, Open-label Study to Evaluate the Safety and Efficacy of VGT-309, a Tumor-Targeted, Activatable Fluorescent Imaging Agent, to Identify Cancer in Subjects Undergoing Lung Cancer Surgery
Brief Title: Phase 2 Study of VGT-309 in Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vergent Bioscience, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGT-309-2-2021USA; 1R44CA277890-01 (NIH)
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: All subjects to be dosed at the same dose level. This is open label and no randomization is required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.32mg/kg VGT-309 (Experimental): Single arm in an open label study
  Interventions: Drug: VGT-309

INTERVENTIONS:
Drug: VGT-309 — VGT-309 is an tumor-targeted, activatable fluorescent imaging agent which will be used with near infrared imaging during surgery to identify tumor.

SUMMARY:
A Phase 2 open label study to evaluate safety and efficacy of VGT-309 to identify cancer in up to 40 subjects undergoing lung cancer surgery.

DETAILED DESCRIPTION:
A Phase 2, open-label study to evaluate the safety and efficacy of VGT-309, a tumor-targeted, activatable fluorescent imaging agent, to identify cancer in subjects undergoing lung cancer surgery. A total of 40 subjects will be enrolled to ensure at least 38 evaluable subjects with the option to expand enrollment by protocol amendment if deemed necessary to meet primary and/or secondary objectives.

Following agreement with and signing of the informed consent, subjects will undergo screening measurements for the study. Assessments include the following, unless they have been done within 4 weeks prior to the anticipated dosing:

1. Medical, surgical and medication history.
2. Complete physical exam, including vital signs and weight.
3. Standard pre-operative chemistry, hematology, coagulation and urinalysis clinical laboratory studies.
4. 12-lead ECG.
5. Serum pregnancy test for females of child-bearing potential.

Following clearance of all enrollment criteria, each subject will receive an IV administration of 0.32 mg/kg VGT-309 at 12-36 hours prior to surgery (refer to section VGT-309 Dosing, below). Upon dosing, subjects will be observed for up to 2 hours and asked about possible treatment emergent adverse events.

Subjects will undergo surgical resection as planned and within the time specified following VGT-309 dosing. Measurements of efficacy will be taken during surgery and during the pathological examination of all surgical specimens.

Following surgery, subjects will be monitored for safety during their hospitalization. After discharge from the hospital, and approximately 14 days post-surgery, the subjects will be contacted by telephone to assess their well-being. Between 19 to 39 days post-surgery, subjects will either return to the clinic or participate in a telehealth visit for final safety assessments. If there are no adverse events requiring further follow up, subjects will then be released from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to sign the informed consent and comply with study procedures.
2. Be between the ages of 18 and 85, inclusive.
3. Be male or female and meet the following conditions:

   1. Female participants must be of non-childbearing potential, or,
   2. If of childbearing potential be non-pregnant or non-lactating and agree to use highly effective contraception from screening through Day 30.
   3. Male participants, if not surgically sterilized, and if engaging in sexual intercourse with a female partner of childbearing potential, must be willing to use highly effective contraception from screening through 30 days post-dose and agree not to donate semen during this waiting period.
   4. Highly effective contraception involves the use of a condom for the male, plus one of the following for the female:

      * Oral, injectable, implantable, intravaginal, or transdermal hormonal contraceptives, or
      * Intrauterine device or intrauterine hormone-releasing system
      * NOTE: Participants who abstain from heterosexual intercourse as their usual and preferred lifestyle, will not be required to use contraception as described above.

   They are required to maintain abstinence from screening through Day 30.
4. Have a lung nodule or mass that might be considered primary lung cancer or lung metastases, whether or not it is biopsy-proven.
5. Be scheduled to undergo standard of care surgical resection for a lung nodule or mass with diagnostic and/or curative intent and meet all pre-operative surgical and anesthesia acceptance criteria.
6. Have acceptable kidney and liver functions at study entry as evidenced by:

   1. Alanine Aminotransferase/Aspartate Aminotransferase (ALT/AST) < 1.5 times the upper limit of normal
   2. Serum creatinine < 1.5 times the upper limit of normal
7. Have an Eastern Cooperative Oncology Group (ECOG) score of 0-2.
8. Meet all standard surgical and general anesthesia requirements.
9. Have not participated in a clinical trial within the last 30 days.

Exclusion Criteria:

1. They are not a candidate for standard of care surgery based on opinion of the surgeon, anesthesiologist, or other consulting physician.
2. They have a known allergy or reaction to indocyanine green (ICG), other radiographic contrast agent, or any component of VGT-309.
3. Have congenital long QT syndrome or QTcF > 450ms (males) or >470ms (females) by history or at Screening ECG.
4. They are prisoners, institutionalized individuals, or are unable to consent for themselves.
5. Have any other co-morbidity or habit that the Investigator believes will interfere with their ability to comply with and complete the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curt Scribner, MD, Study Director — Vergent Bioscience
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- VGT-309: VGT-309 0.32mg/kg IV 12-36 hours pre surgery
Period: Overall Study
Arm/Group | VGT-309
Started | 40
Dosing | 40
Surgery | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One-time dose by IV infusion over 15-20 minutes using a syringe pump between 12-36 hours prior to the start of surgery
Groups:
- VGT-309 0.32mg/kg: One-time dose by IV infusion over 15-20 minutes using a syringe pump between 12-36 hours prior to the start of surgery
Arm/Group | VGT-309 0.32mg/kg
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 27
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 66 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 29
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 40
Height [Mean (Standard Deviation); unit: cm] | 165.33 (13.863)
Weight [Mean (Standard Deviation); unit: kg] | 77.61 (23.658)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.62 (9.349)

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Event (CSE)
Description: Identification of the proportion of subjects with at least one CSE as defined by:
  A. Localization of a Pulmonary Nodule using VGT-309 near-infrared (NIR) Imaging when white light and palpation failed to identify a nodule.
  B. Synchronous Lesion Identification using VGT-309 NIR Imaging when not identified by white light and palpation.
  C. Positive Margin Identification with only VGT-309 NIR Imaging when deemed negative by the surgeon by white light and palpation.
Time Frame: Day of surgery
Population: Efficacy Population: All subjects who received any amount of VGT-309 and had surgery with NIR imaging
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Groups:
- VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery: Subjects who received VGT-309 and underwent intraoperative NIR imaging.
Arm/Group | VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery
Number analyzed (Participants) | 40
Proportion of subjects | 0.425 [0.270 to 0.591]
Statistical Analysis 1: Comparison: VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery; Single arm open-label; Test type: Other — Summary statistics of quantitative data, one-sided exact binomial test for null hypothesis, Clopper-Pearson method for 95% exact confidence intervals; p < .0001, Exact Binomial Test; Proportion = 0.425, 95% CI 2-sided [0.270 to 0.591] — The Parameter Dispersion Value is the asymptotic standard error of the proportion

2. Secondary Outcome: Sensitivity
Description: Sensitivity is defined as the probability that tissue fluoresces intraoperatively when it is cancer as confirmed by histology.
  Sensitivity = (True Positive)/(True Positive + False Negative)
Time Frame: Day of surgery
Measure: Number (95% Confidence Interval); unit: Proportion of lesions
Units Other Than Participants: lesions
Arm/Group | VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery
Number analyzed (Participants) | 40
Number analyzed (lesions) | 55
Proportion of lesions | 0.850 [0.675 to 0.939]
Statistical Analysis 1: Comparison: VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery; Test type: Other; Proportion = 0.850, 95% CI 2-sided [0.675 to 0.939]

3. Secondary Outcome: Negative Predictive Value
Description: Negative predictive value is defined as the probability that a tissue sample does not contain cancer on histologic exam if it does not fluoresce intraoperatively.
  Negative Predictive Value = (True Negative)/(True Negative + False Negative)
Time Frame: Day of surgery
Population: Efficacy Population: All subjects who received any amount of VGT-309 and had surgery with NIR imaging
Measure: Number (95% Confidence Interval); unit: Proportion of lesions
Units Other Than Participants: lesions
Arm/Group | VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery
Number analyzed (Participants) | 40
Number analyzed (lesions) | 55
Proportion of lesions | 0.455 [0.202 to 0.733]
Statistical Analysis 1: Comparison: VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery; Test type: Other; Proportion = 0.455, 95% CI 2-sided [0.202 to 0.733]

4. Secondary Outcome: Specificity
Description: Specificity is defined as the probability that tissue does not fluoresce intraoperatively when it is not cancerous as confirmed by histology.
  Specificity = (True Negative)/(True Negative + False Positive)
Time Frame: Day of surgery
Population: Efficacy Population: All subjects who received any amount of VGT-309 and had surgery with NIR imaging
Measure: Number (95% Confidence Interval); unit: Proportion of lesions
Units Other Than Participants: lesions
Arm/Group | VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery
Number analyzed (Participants) | 40
Number analyzed (lesions) | 55
Proportion of lesions | 0.333 [0.126 to 0.633]
Statistical Analysis 1: Comparison: VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery; Test type: Other; Proportion = 0.333, 95% CI 2-sided [0.126 to 0.633]

5. Secondary Outcome: Positive Predictive Value
Description: Positive predictive value is defined as the probability that a tissue sample contains cancer on histologic exam if it fluoresces intraoperatively.
  Positive Predictive Value = (True Positive)/(True Positive + False Positive)
Time Frame: Day of surgery
Population: Efficacy Population: All subjects who received any amount of VGT-309 and had surgery with NIR imaging
Measure: Number (95% Confidence Interval); unit: Proportion of lesions
Units Other Than Participants: lesions
Arm/Group | VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery
Number analyzed (Participants) | 40
Number analyzed (lesions) | 55
Proportion of lesions | 0.773 [0.650 to 0.862]
Statistical Analysis 1: Comparison: VGT-309 0.32mg/kg IV Given 12-36 Hours Prior to Surgery; Test type: Other; Proportion = 0.773, 95% CI 2-sided [0.650 to 0.862]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of dosing through completion of the End-of-Study Visit (Days 22-36)
Description: ClinicalTrials.gov definition of "Adverse Events" was used for data collection and reporting
Arm/Group | VGT-309 0.32mg/kg
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 8/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VGT-309 0.32mg/kg (N=40)
Ileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VGT-309 0.32mg/kg (N=40)
Procedural pain (Injury, poisoning and procedural complications) | 40
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 17
Hypertension (Vascular disorders) | 2
Sinus bradycardia (Cardiac disorders) | 6
Supraventricular extrasystoles (Cardiac disorders) | 4
Supraventricular tachycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Aspartate aminotransferase increased (Investigations) | 4
Amylase increased (Investigations) | 2
Gamma-glutamyl transferase increased (Investigations) | 2
Urinary retention (Renal and urinary disorders) | 7
Fatigue (General disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Hallucination (Psychiatric disorders) | 2
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT05400226/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT05400226/SAP_001.pdf